CLINICAL TRIAL: NCT03502525
Title: Break the Cycle: Adapting Break the Cycle to Reduce Initiation Into Injecting Drug Use in Tallinn, Estonia and New York City, USA
Brief Title: Break the Cycle: Prevention for Reducing Initiation Into Injection Drug Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: University of Tartu (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GCO 15-1445; 5DP1DA039542-05 (NIH)
Record Dates: First submitted 2018-04-11; First posted 2018-04-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2020-02

CONDITIONS: Substance Abuse, Intravenous; Prevention and Control
MeSH Terms: conditions — Substance Abuse, Intravenous

STUDY DESIGN:
Intervention Model Description: In the second and third iterations of the study in New York City, participants are randomized to either Break the Cycle or an attention control intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Break the Cycle Intervention (Experimental): Break the Cycle intervention uses motivational interviewing to enhance current injectors' motivation and skills to avoid helping with and promoting first injections among non-PWID.
  Interventions: Behavioral: Break the Cycle Intervention
- Bacterial Infection Prevention (Active Comparator): Bacterial Infection Prevention is an attention control intervention. The content of Bacterial Infection Prevention is representative of the infection prevention information injection drug users ought to receive, and sometimes do, when they engage with service providers, such as syringe exchange programs. Bacterial Infection Prevention does not use Motivational Interviewing principles, but is more informational/educational in nature. This intervention focuses on bacterial infection risks that accompany injection drug use, with a special focus on risk reduction, identification, and treatment of abscesses and endocarditis.
  Interventions: Behavioral: Bacterial Infection Prevention

INTERVENTIONS:
Behavioral: Break the Cycle Intervention — The intervention uses motivational interviewing to enhance persons who inject drugs' (PWID) motivation and skills to avoid helping non-PWID transition to injecting. The intervention entails discussions with participants in 8 areas: the participant's first time injecting; the participant's exposures to situations where helping with non-PWIDs' first injections is an option, and the extent to which they helped; their behaviors that might encourage non-PWID to inject for the first time; the risks associated with injection drug use; role-playing in which participants develop behaviors and scripts for avoiding or refusing requests to initiate non-PWID into injection; role- playing talking with other PWID about not encouraging non-PWID to start injecting; imparting safer injection practices when helping with a first injection seems like the best option; and receiving training in and using naloxone to reverse overdoses.
  Arms: Break the Cycle Intervention
Behavioral: Bacterial Infection Prevention — Bacterial Infection Prevention is an attention control intervention. The content of Bacterial Infection Prevention is representative of the infection prevention information injection drug users ought to receive, and sometimes do, when they engage with service providers, such as syringe exchange programs. Bacterial Infection Prevention does not use Motivational Interviewing principles, but is more informational/educational in nature. This intervention focuses on bacterial infection risks that accompany injection drug use, with a special focus on risk reduction, identification, and treatment of abscesses and endocarditis.
  Arms: Bacterial Infection Prevention

SUMMARY:
Break the Cycle is a two-session, one-on-one, in-person intervention study designed to reduce the role persons who inject drugs (PWID) play initiating non-PWID into injection drug use. Study implementation is at two sites: New York City and Tallinn, Estonia. At baseline, quantitative data are collected via a structured computer-assisted personal interview, after which the intervention is conducted. At the 6-month follow-up, a modified version of the interview is repeated.

In Tallinn, and in it's first iteration in NYC, Break the Cycle used a pre- versus post- design to compare the proportion of participants who helped with first injections, and who promoted injecting among non-PWID, in the 6 months prior to baseline with the proportions at the 6-month follow-up. Based on previous research on the intervention and on the underlying theory of motivational interviewing, increases in helping and promoting behaviors between baseline and follow-up would indicate that the intervention was not effective regardless of their effect size. Accordingly, the hypotheses that the intervention will produce reductions in assisting with first injections and engaging in injection promoting behaviors will be evaluated using one-tailed statistical tests. Break the Cycle intervention follows a motivational interviewing approach to enhance current injectors' motivation and skills to avoid helping with and promoting first injections among non-PWID. The intervention's core is a discussion between an interventionist and each participant on the following eight topics: the participant's first time injecting drugs; the participant's exposures to situations where helping with others' first injections is an option, and the extent to which they have helped; PWIDs' behaviors that might encourage non-PWID to inject for the first time; the range of risks associated with injection drug use; role-playing scenarios in which the participant develops behaviors and scripts for avoiding or refusing requests to initiate others into injection drug use; role- playing talking with other PWID about not encouraging non-PWID to start injecting; imparting safer injection practices when helping with a first injection seems like the best option; and receiving training in and using Narcan to reverse overdoses.

In the second iteration of Break the Cycle in New York City, a second arm to the trial was added: an attentional control intervention, Bacterial Infection Prevention. The content of Bacterial Infection Prevention is representative of the infection prevention information injection drug users ought to receive, and sometimes do, when they engage with service providers, such as syringe exchange programs. Bacterial Infection Prevention does not use Motivational Interviewing principles, but is more informational/educational in nature. This intervention focuses on bacterial infection risks that accompany injection drug use, with a special focus on risk reduction, identification, and treatment of abscesses and endocarditis. Participants eligible for Break the Cycle are randomized to either receive the Break the Cycle intervention or the Bacterial Infection Prevention intervention. Enrollment in this iteration ended in March 2020, with the advent of the Covid pandemic in the United States.

The third iteration of the Break the Cycle intervention in New York City will transform the second iteration into a phone-based study in which both Break the Cycle and Bacterial Infection Prevention are delivered to participants over the telephone. Both interventions have been slightly abbreviated to adjust to phone delivery. This iteration will commence in early spring, 2021.

ELIGIBILITY:
Inclusion Criteria:

* have injected drugs non-medically in the last 2 months
* able to provide informed consent
* age 18 or older
* able to participate in the interview and intervention in English (in New York City), Russian or Estonian (in Tallinn, Estonia)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Number of participants helping with first injections | 6 months
  Number of participants who helped persons who do not inject drugs with a first injection

SECONDARY OUTCOMES:
Number of participants who say positive things | 6 months
  Number of participants who saying positive things about injecting to persons who do not inject drugs
Number of participants injecting in front of other people | 6 months
  Number of participants injecting in front of people who do not inject drugs
Number of participants offering to give first injection | 6 months
  Number of participants offering to give a first injection to persons who do not inject drugs

CONTACTS AND LOCATIONS:
Overall Officials: Don Des Jarlais, PhD, Principal Investigator — New York University; Anneli Uuskula, PhD, Principal Investigator — University of Tartu
Locations (2):
- New York University, New York, New York, United States
- University of Tartu, Tallinn, Estonia

IPD SHARING:
Plan to Share IPD: No